CLINICAL TRIAL: NCT03551847
Title: The Effect of Oral Antibiotics on Synovial Fluid Leukocyte Count and Differential for the Diagnosis of Periprosthetic Hip and Knee Infection
Brief Title: The Effect of Oral Antibiotics on Synovial Fluid and Differential for the Diagnosis of Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll any subjects, closed study
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16071701
Record Dates: First submitted 2017-10-26; First posted 2018-06-11 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral antibiotic therapy group (Experimental): This group will receive preoperative oral antibiotic therapy tailored to the infecting organism (if identified) for two weeks before the time of revision surgery
  Interventions: Drug: Antibiotic
- No antibiotic therapy group (Active Comparator): This group will not receive preoperative oral antibiotic therapy.
  Interventions: Drug: No antibiotics

INTERVENTIONS:
Drug: Antibiotic — The intervention involves giving an infected patient antibiotics.
  Arms: Oral antibiotic therapy group
Drug: No antibiotics — The intervention involves not giving an infected patient antibiotics.
  Arms: No antibiotic therapy group

SUMMARY:
Periprosthetic joint infection following total hip or knee arthroplasty is a rare but potentially devastating complication. Accurate diagnosis of these infections remains one of the most challenging undertakings in orthopaedics. Multiple studies have shown the high diagnostic accuracy of synovial fluid white blood cell count (WBC) and neutrophil percentage (%PMNs) in detecting PJI. This study's goal is to evaluate how antibiotics affect those two important diagnostic measures.

DETAILED DESCRIPTION:
Periprosthetic joint infection (PJI) following total hip or knee arthroplasty is a rare but potentially devastating complication. Accurate diagnosis of these infections remains one of the most challenging undertakings in orthopaedics. Clinical presentation of PJI may be subtle and distinguishing between infection versus aseptic issues can be difficult. Currently no diagnostic approach has been developed that accurately and unequivocally diagnoses PJI.

Multiple studies have shown the high diagnostic accuracy of synovial fluid white blood cell count (WBC) and neutrophil percentage (%PMNs) in detecting PJI. This has led to incorporation of these two parameters into criteria for the diagnosis of PJI. WBC and %PMN cutoffs have been published for prosthetic hips and knees in both the acute and chronic setting. Meanwhile, synovial fluid cell counts are believed to be of particular value when patients present on systemic antibiotics, which have been shown to compromise intraarticular cultures by causing false negative results.

However, the effect of antibiotics on synovial fluid cell count and differential has not been well delineated. One prospective study by Trampuz et al. of 133 synovial fluid specimens prior to total knee revisions noted that patients receiving antimicrobial agents had lower leukocyte counts than did those who were not receiving antimicrobial agents. To the contrary, a recent animal study examined intra-articular administration of the antibiotic amikacin in horses and reported a statistically significant increase in the synovial nucleated cell count. The effect of antibiotics on synovial fluid WBC and %PMN thus remains unclear.

Furthermore, to reduce false-negative culture results, it is recommended that patients be off of antibiotics for a minimum of two weeks prior to obtaining samples for culture. Investigators have shown reduced false-negative culture rates in patients not taking antibiotics prior to surgery compared to those taking antibiotics at the time of surgery. However, the two-week time interval is relatively arbitrary and adequate supporting data do not exist.

The primary aim of this study is to evaluate how antibiotics affect synovial fluid leukocyte and differential counts. A secondary aim is to assess how long patients need to be off of antibiotic therapy to generate accurate synovial fluid cultures. Further examination of the effects of systemic antibiotics on synovial fluid composition will provide valuable information for clinicians caring for patients with possible PJI.

ELIGIBILITY:
Inclusion Criteria:

1. Patient>18 years old.
2. Patient with a prosthetic hip or knee in place.
3. Patient with PJI of the hip or knee based on MSIS criteria3(Table 1).
4. Patient off of antibiotics for a minimum of two weeks prior to preoperative joint aspiration.
5. Patient with a culture-positive preoperative joint aspiration

Exclusion Criteria:

1. Inadequate preoperative or intraoperative synovial fluid sample to perform synovial fluid WBC, %PMN and aerobic/anaerobic cultures.
2. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
A change in synovial fluid white blood cell count with antibiotic treatment | pre-operative to intraoperative
  White blood cell count will be measured from synovial fluid. This fluid will be sent to our in-house laboratory testing facility. WBC is measured as the total number per mL of fluid.
A change in synovial fluid neutrophil percentage with antibiotic treatment | pre-operative to intraoperative
  Neutrophil percentage will be measured from synovial fluid. This fluid will be sent to our in-house laboratory testing facility. %PMN is a percentage out of total white blood cell count.

SECONDARY OUTCOMES:
A change in culture results with antibiotic treatment | pre-operative to intraoperative
  Synovial fluid will be sent to our in-house lab and they will try and grow cultures from this fluid to see if they can identify the organism causing the infection.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Professor of Orthopaedic Surgery
Locations (1):
- Rush University medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No